CLINICAL TRIAL: NCT06426849
Title: Effects of Liuzijue Exercise Versus Tai Chi Chuan Exercise in Improving Dyspnea Index and Pulmonary Function in Patients With Asthma
Brief Title: Effects of Liuzijue Exercise Versus Tai Chi Chuan Exercise in Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rec/01815 Maria Akbar
Record Dates: First submitted 2024-05-19; First posted 2024-05-23 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Asthma
Keywords: Liuzijue exercise; Tai Chi Chuan exercise; Dyspnea Index; Pulmonary Function; Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP A (Experimental): LiuzijueExercise will be performed by delivering 6 distinct sounds,("xū", "hē", "hū", "sī", "chuī", and "xī") through termination along with comparing body activities.
  Interventions: Other: Liuzijue Exercise
- GROUP B (Experimental): 10 FORM OF YANG NG STYLE Tai Chi Chuan Exercise that combines deep diaphragmatic breathing and relaxation with many fundamental postures.
  Interventions: Other: Tai Chi Chuan Exercise

INTERVENTIONS:
Other: Liuzijue Exercise — LiuzijueExercise includes inhalation and exhalation through various mouth patterns to manage and control the rise and fall of the breath in the body. It is performed by delivering 6 distinct sounds, (xū,hē, hū sī, chuī, and xī) through termination along with comparing body activities.
  The following are 6-8 vital parts of body movements:
  1. Swaying and twisting
  2. Hip rotations
  3. Arm movements
  4. Knee bends
  5. Foot pivots
  6. Spine elongation
  7. Hand gestures
  8. Breath synchronization Frequency: 1 session per day for a week Intensity:In first week 1 set of Luizijue exercise will be performed then progressively increase to 4 sets till 6th week .
  Total Time for Session; 40 minutes Warm-up Time: 10 minutes with pursed lip breathing Cool Down Time: 10 minutes with upper body gentle stretching. Exercise Duration: 20 minutes for Luizijue Exercise.
  Arms: GROUP A
Other: Tai Chi Chuan Exercise — Tai Chi Chuan Exercise combines deep diaphragmatic breathing and relaxation with many fundamental postures.
  Names of the 10 Movements in Sequence
  1. Commencing Form
  2. Repulsing the Monkey
  3. Brush Knee
  4. Parting the Horse's Mane
  5. Cloud Hands
  6. Golden Cockerel Standing on the Left, then the Right
  7. Kick Out Right, Kick Out Left
  8. Grasping the Bird's Tail
  9. Cross Hands or Embrace the Tiger
  10. Closing Form Frequency: 3 sessions / week Intensity: Initially each posture will be performed 3 times then progressively leads to 6 or 10 reps according to patient tolorance.
  Total Time for Session; 40 minutes Warm-up Time: 10 minutes with pursed lip breathing Cool Down Time: 10 minutes with upper body gentle stretching. Exercise Duration: 20 minutes for Tai Chi Chuan Exercise.
  Arms: GROUP B

SUMMARY:
To analyze either Liuzijue exercise or Tai Chi Chuan exercise is effective in improving dyspnea index and pulmonary function in patients with asthma. In the general population, the rate of asthma is increasing day by day because of environmental and occupational risk factors which is becoming a burden. It causes shortness of breath, decreases lung volume, and disturbs quality of life. This study aims to improve dyspnea index, lung volume and quality of life of the patients with asthma.

DETAILED DESCRIPTION:
Liuzijue Exercise is the most popular exercise in ancient Chinese literature which is compiled by the Chinese Qigong Management Centre. Liuzijue exercise includes inhalation and exhalation through various mouth patterns to manage and control the rise and fall of the breath in the body. It is performed by delivering 6 distinct sounds, ("xū", "hē", "hū", "sī", "chuī", and "xī") through termination along with comparing body activities. It is very helpful to improve pulmonary functions, exercise capacity, and quality of life of patients with pulmonary disease.

Liuzijue exercise takes on the backward abdominal breathing technique joined with physical exercises, which can practice the diaphragm and chest auxiliary respiratory muscles. Hence, the patient's breathing time is extended, and the breathing profundity increments. To accomplish the reason for expanding the gas exchange rate of the lungs and enhancing the lung capacity. Tai Chi Chuan is a traditional Chinese Exercise that is significant in improving the pulmonary functions of asthmatic patients.

Tai Chi (10 forms of yang style ) significantly improves the exercise capacity of patients with lung disease. Tai Chi seems to have physiologic and psychosocial benefits and appears to be protected and viable in advancing balance control, adaptability, and cardiovascular fitness for older adults.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed case of Asthma for last 6 months
* Patients with mild to moderate asthma
* On spirometry FEV1/FVC ratio less than 70%
* MRC- Grade 2 and 3

Exclusion Criteria:

* Refusal to consent.
* Unstable vitals.
* Diagnosed with any lung disease.
* Uncontrolled Hypertension.
* Diagnosed Tumor.
* Patient with Stroke and other neurological conditions.
* Patient with active Tuberculosis or other infectious disease.
* Patients with history of heart failure or any other cardiovascular condition

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Dyspnea index | 6 weeks
  From baseline till 2nd, 4th, and 6th week measured throug Modified Medical Research Council (mMRC) dyspnoea scale. It is a self-rating scale to quantify the level of incapacity that breathlessness presents on everyday activity on a scale from Grade 0 to 4.
  Grade 0: No shortness of breath besides on exhausting activity Grade1: Breathlessness while hustling fair and square or strolling along a slight slope Grade 2: Strolls more slow than individuals of same age fair and square in light of shortness of breath or needs to stop to take breath while strolling at their own speed fair and square Grade 3: Stop for breath subsequent to strolling ∼100 m or following couple of moments fair and square.
  Grade 4: Excessively breathless to take off from the house, or breathless while dressing or stripping down
Forced Expiratory Volume in 1 second (FEV1) | 6 weeks
  Changes from the Baseline, the digital spirometer is used in the clinical setting to analyze

SECONDARY OUTCOMES:
Asthma Quality of life | 6 Weeks
  From baseline till 6th week measured through Asthma Control Questionnaire that individuals answer in regards to the recurrence of asthma symptoms over 6 weeks.
  Each answer has a numeric value. The asthmatic individual adds their score to decide their degree of asthma symptoms control. Score ranges from 5 to 25. A score 20 to 25 indicate well controlled asthma while score ranges between 5 to 6 indicated poor controlled asthma.

CONTACTS AND LOCATIONS:
Overall Officials: Mehwish Waseem, MSPT-CPPT, Principal Investigator — Riphah International University
Locations (1):
- Tehsil Headquarter Hospital, Chichawatni, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No